CLINICAL TRIAL: NCT02606851
Title: China Survey of Proton Pump Inhibitor Empirical Treatment in Management of Outpatients With Gastroesophageal Reflux Disease
Brief Title: Proton Pump Inhibitor Empirical Treatment in Management of Outpatients With Gastroesophageal Reflux Disease.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1844R00002
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Patients With Typical Symptoms of GERD (GERD Q >= 8)
Keywords: Proton Pump Inhibitor, GERD, GERD Q
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
China Survey of Proton Pump Inhibitor Empirical Treatment in Management of Outpatients with Gastroesophageal Reflux Disease

DETAILED DESCRIPTION:
To estimate the overall responder rate after 4 weeks of Proton Pump Inhibitor empirical treatment This will be a multicenter prospective observational study carried out in China. Investigator will collect data in a pre-specified Case Report Form from the outpatient. Informed consents will be needed. Investigator will provide patient diary card to each patient for them to note down the symptom frequency every day. Main data from each outpatient will include demographics, Gerd Q, symptom frequency and Proton Pump Inhibitor empirical treatment. Data from each outpatient will be collected on the screening day, 2 weeks and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, and any race, Age ≥ 18 years and≤ 65 outpatients.
* Gastroenterologists already prescribe PPI standard dose bid as empirical treatment.
* GerdQ≥8
* The subject will not have endoscopy within 4 weeks after enrolment.
* Ability to provide informed consent, adhere to the study visit schedule, and complete all study assessments and complete the patient diary by his/herself.

Exclusion Criteria:

* If participating in any interventional clinical trial.
* Patient with alarm symptom of oncology(weight loss, recurrent dysphagia, anemia, hematemesis, melena).
* Continuous application of nonsteroidal anti-inflammation drugs or acid suppressive drug within 2 weeks before screening.
* The need for H2-receptor antagonists (H2RA) including cimetidine, ranitidine and famotidine or sucralfate, antacids, traditional Chinese medicine and prokinetics during the upcoming 4 weeks (study duration).
* Previous gastroesophageal surgery.
* Upper gastrointestinal malignancy, achalasia, and esophageal spasm or stricture.
* Peptic ulcer
* Diabetes
* Cerebral vascular disease
* Zollinger-Ellison syndrome
* Scleroderma
* Hiatus hernia women
* Pregnant or lactating women
* Any other subjects were not suitable to this study in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population that will be included in the NIS are the consecutive outpatients between 18 and 65 years old with Gerd Q ≥ 8, who will not have endoscopy within 4 weeks while gastroenterologists already prescribe PPI as empirical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
The overall responder rate | After 4 weeks of Proton Pump Inhibitor empirical treatment
  The overall responder rate after 4 weeks of Proton Pump Inhibitor empirical treatment. Responder is defined as heartburn/regurgitation frequency ≤1 days during 7 days before evaluation visit, assessed using Gerd Q questionnaire at each post-baseline visit.

SECONDARY OUTCOMES:
The overall responder rate | After 2 weeks of Proton Pump Inhibitor empirical treatment
  The overall responder rate after 2 weeks of Proton Pump Inhibitor empirical treatment
The proportion of patients in each Gerd Q cut-off range at each visit | At each visit (baseline, 2 weeks and 4 weeks)
  The proportion of patients in each Gerd Q cut-off range at each visit (Gerd Q range: ≤2; 3-7; 8-10; 11-18)
The responder rate of different Proton Pump Inhibitor empirical treatment | After 2 and 4 weeks of different PPIs empirical treatment
  The responder rate respectively after 2 and 4 weeks of different Proton Pump Inhibitor empirical treatment
The median time to response overall and for different Proton Pump Inhibitor, respectively | During 4 weeks of whole study
  The median time to response (heartburn/regurgitation frequency ≤1 days during last 7 days assessed using patient's diary card) overall and for different Proton Pump Inhibitor, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Duowu Zou, leading PI, Principal Investigator — Changhai Hospital
Locations (10):
- China (10):
  - Research Site, Beijing
  - Research Site, Benijin
  - Research Site, Changchun
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Xining

REFERENCES:
- See also: GID1844R00002 CSR-Synopsis_final 1 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3946&filename=GID1844R00002_CSR-Synopsis_final_1.pdf